CLINICAL TRIAL: NCT05541848
Title: Clinical Benefits of a Multimodal Physiotherapy Programme in Fighter Pilots With Flight-related Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carlos Fernández-Morales, Principal Investigator, Universidad de Extremadura
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 03
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Neck Pain
Keywords: fighter pilots; flight-related neck pain; disability; electric massage; Therapeutic exercise
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in the control group will not receive any intervention and will continue with their normal combat and flight exercise activities. They will be asked not to take medication or seek alternative treatments.
- Experimental group (Experimental): Participants in the experimental group will follow a supervised ELGF program. Subsequently, they will receive an intervention based on manual therapy combined with electrical stimulation called electro-massage.
  Interventions: Other: Cervical supervised exercises with laser-guided feedback (ELGF); Other: Interferential current electro massage (ICE)

INTERVENTIONS:
Other: Cervical supervised exercises with laser-guided feedback (ELGF) — Cervical supervised exercises with laser-guided feedback (ELGF) is defined as a procedure of proprioceptive training based on a type of therapeutic exercise that provides external feedback to exercise, achieving an improvement in range of motion and postural control in subjects with spinal pain. For the performance of the exercise program, "Motion Guidance Clinician Kit" (Motion Guidance LLC, Denver, CO, USA.) was used. The program consisted of 4 exercises, which progressed in difficulty according to the tolerance achieved over the course of the sessions: a) Maintaining the head position (cervical stabilisation); b) Cervical flexion-extension; c) Right-left rotations; d) Right-left lateral-flexions. Each exercise consisted of 4 series of 8 repetitions, except the first one, in which the head position is maintained by pointing the laser at the centre of the panel for 30 seconds (4 series). The average time to complete the entire program did not exceed 14 minutes.
  Arms: Experimental group
Other: Interferential current electro massage (ICE) — Interferential current electro-massage (ICE) is defined as a technique which combines simultaneously manual therapy (massage) and ICT. We used a current bipolar mode, using a carrier frequency of 4000 Hz at constant voltage and an amplitude-modulated frequency of 100 Hz (Sonopuls 692®; Enraf-Nonius BV, Rotterdam, The Netherlands), was administered. The intensity was set to provide a strong and comfortable tingling, without evoking muscle twitches even though a slight vibration (fasciculation) was allowed. The sequence combined (A) superficial stroke over the neck-shoulder for 30-45 seconds; (B) deep sliding movements, alone or (C) combined with shoulder drop, for 4-5 minutes; (D) bilateral kneading of the upper trapezius (4-5 minutes); (E) slight stretching of cervical muscles (upper trapezius, sternocleidomastoid, and levator scapulae); and repetition of step (A). The electro-massage protocol lasted 15 minutes.
  Arms: Experimental group

SUMMARY:
The aim of this study was to analyse the immediate effects of a 4-week multimodal physiotherapy program which combines cervical supervised exercises with laser-guided feedback (ELGF) and interferential current electro massage (ICE) in fighter pilots with flight-related neck pain.

DETAILED DESCRIPTION:
Flight-related neck pain constitutes a clinical entity related to the performance and flight safety of fighter pilots. The aim of this study was to analyse the effectiveness of a multimodal physiotherapy program which combines supervised Exercise with Laser-Guided Feedback (ELGF) and Interferential Current Electro-Massage (ICE) in fighter pilots with flight-related neck pain.

31 pilots were randomly allocated into two groups (Experimental Group n=14; Control Group n = 17). The intervention consisted of 8 sessions (twice a week) for 4 weeks. As primary outcome measures the following variables were measured: perceived pain intensity (Numeric Pain Rating Scale) and neck disability (Neck Disability Index). The secondary outcome measures were: cervical range of movement (CRoM), joint position sense error (JPSE) and pressure pain threshold (PPT).

ELIGIBILITY:
Inclusion Criteria:

* Flight pilots (male and female) who, at the time of the assessment, were an instructor or student attached to the 23th Wing of Talavera Air Base, Spanish Air Force (SAF), Badajoz.
* Flight pilots diagnosed with flight-related neck pain according to the International Classification proposed by an expert panel of the North Atlantic Treaty Organisation (NATO).
* A minimum perceived pain of 3/10 on the Visual Analogue Scale (VAS) in the early-morning assessment.
* Scores of ≥5 points on the Neck Disability Index (NDI), and a cervical-repositioning error of ≥4.5°.

Exclusion Criteria:

* Cervical pain with radiation to the upper limbs and/or radiculopathy.
* Cervical spine surgery with or without the presence of a metal implant.
* Having received physiotherapy or any other routine medical care six weeks prior to data collection.
* Being involved in ongoing medical-legal conflicts.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4 weeks.
  Numeric Pain Rating Scale (NPRS) is a 11-point numeric rating scale, where 0 denotes "no pain" and 10 denotes "the maximum bearable pain". The minimum clinically important difference (MCID) for this tool has been established at 1.5 points and the minimum detectable change (MDC) at 2.6 points, in individuals with neck pain. The NPRS is a valid scale with moderate test-retest reliability in this population (Intraclass Coefficient Correlation (ICC): 0.76, 95% CI 0.58 to 0.93).
Cervical Joint Position Sense Error (JPSE) | 4 weeks.
  This test consists of a visual measurement of the error in moving the head to the initial neutral position after active cervical rotation.

SECONDARY OUTCOMES:
Cervical Range of Motion (CRoM) | 4 weeks.
  For the evaluation of CROM, a conventional EnrafNonius® two-branch goniometer was used. Subjects were placed in a seated position on a stool, with a neutral neck and head position. The range of active cervical mobility presented by the patients was measured in reference to the three planes of the space. In the sagittal plane, the degrees of mobility to flexion and extension were measured, in the frontal plane the right and left inclinations, and in the transverse plane both rotations.
Pressure Pain Threshold (PPT) | 4 weeks.
  A mechanical pressure Fisher algometer (Force Dial model FDK 40) with a 1 cm² area contact head was used to measure the pressure pain threshold. The reliability of pressure algometry has been found to be high [intraclass correlation coefficient = 0.91 (95% confidence interval, 0.82-0.97)]. With the participant in supine, the pressure pain threshold of the the myofascial trigger point nº2 of the upper trapezius muscle according to Travell and Simons and the central trigger point of the sternocleidomastoid muscle was bilaterally evaluated. Also, in sitting position the pressure pain threshold of the myofascial trigger point of the scapula elevator muscle was bilaterally evaluated. The minimal clinically important difference (MCDI) is 1.2 Kg/cm2.
Standard Deviation 1 (SD1) | 4 weeks.
  It indicates the sensitivity of short-term variability in HRV non-linear spectrum. It is considered an indicator of parasympathetic activity.
Standard Deviation 2 (SD2) | 4 weeks.
  It is a diameter from Poincaré plot which indicates the degree of longitudinal dispersion. It is thought to reflect long-term changes in RR intervals and it is considered an inverse indicator of parasympathetic activity.
Min_HR | 4 weeks.
  Minimum heart rate variability.
Max_HR | 4 weeks.
  Maximum heart rate variability.
Mean_HR | 4 weeks.
  It corresponds to the interval between two beats (R peaks on the ECG).
pNN50 | 4 weeks.
  Percentage of consecutive RR intervals that differ by more than 50 ms from each other. A high value of pNN50 provides valuable information about high spontaneous HR.
Low Frequency Power (LF) | 4 weeks.
  Situated between 0.04 and 0.15 Hz. In long-term recordings it provides us with more information about the activity of the SNS.
High Frequency Power (HF) | 4 weeks.
  They are located between 0.15 and 0.4 Hz. HF is clearly related to PNS activity and has a relaxation-related effect on HR2.
Low/High Frequency ratio (HF/LF) | 4 weeks.
  From low frequency and high frequency ratio of the HRV spectral analysis result we can estimate the vagal (related to relaxation and HF) and sympathetic (related to stress and LF) influence. Thus we can estimate sympathetic-vagal balance.
Myoelectric activity | 4 weeks.
  The electromyography (EMG) signal of the upper trapezius muscle was recorded during 3 step contractions of shoulder elevation force (15%-30% maximal voluntary contraction). The highest value of the three contractions was taken. The signal of the sternocleidomastoid muscle was recorded during 3 billateraly step contractions of neck flexión and antepulsion neck force. Both contractions were performed in a combined and simultaneous movement, recreating the movement produced by the reaction forces in the takeoff and landing of the fighter jet. Both movements were made at 15%-30% maximal voluntary contraction, as used by Calamita et al on the same musculature in subjects with nonspecific neck pain.
Kinesophobia | 4 weeks.
  The Spanish version of the TSK-11 was used to measure fear of movement. Higher scores indicate greater fear-avoidance behaviors. The TSK-11 has demonstrated acceptable internal consistency and validity.
Catastrophizing Pain | 4 weeks.
  The Pain Catastrophizing Scale (PCS) is a self-administered scale of 13 items and one of the most used to assess catastrophism of pain. The subjects take their past painful experiences as a reference and indicate the degree to which they experienced each of the 13 thoughts or feelings on a 5-point Líkert scale ranging from 0 (never) to 4 (always). The theoretical range of the instrument is between 13 and 62, indicating low scores, little catastrophism, and high values, high catastrophism.
Sympathetic/parasympathetic ratio (S/PS) | 4 weeks.
  S/PS is expressed as the quotient of SS and SD1, and it is considered to reflect autonomic balance - that is, the relationship between sympathetic and parasympathetic activity
Stress Score | 4 weeks.
  It is an index to facilitate physiological interpretation of Poincaré plot. It is expressed as the inverse of the SD2 diameter multiplied by 1000 and is considered directly proportional to the sympathetic activity in the sinus node.
Neck Disability Index (NDI) | 4 weeks.
  The degree of cervical disability involvement was measured through the Neck Disability Index (NDI), translated into Spanish, presenting optimum reliability and internal validity. It consists of 10 sections, 4 of them are related to subjective symptoms and the other 6 are related to basic activities of daily life.
  Each of the sections presents 6 possible responses, scoring these from 0 to 5 according to progression of functional disability.
  Scores less than 5 points indicate non-disability, between 5-14 points indicates mild disability, values between 30-48 points moderate disability, between 50-64 points severe disability and those that exceed 70 points represent complete disability.
Root Mean Square of the Successive Differences (RMSSD) | 4 weeks.
  It indicates the degree of activation of the Parasympathetic Nervous System on the cardiovascular system. It is obtained from the square root of the mean value of the sum of the squared differences of all successive RR intervals. This parameter reports the short-term variations of the RR intervals. It is directly associated with short-term variability.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo-Antúnez, PhD, Study Director — University of Extremadura; Carlos Fernández-Morales, PT, MSc, Principal Investigator — University of Extremadura
Locations (1):
- University of Extremadura, Badajoz, Spain

REFERENCES:
- [Background] Farrel P, Shender B, Goff C, Baudou J, Crowley J, Davies M. 252 HFaMPNRTG. Aircrew Neck Pain Prevention and Management. NATO Reserach and Technology Organisation. 2019;
- [Background] Revel M, Andre-Deshays C, Minguet M. Cervicocephalic kinesthetic sensibility in patients with cervical pain. Arch Phys Med Rehabil. 1991 Apr;72(5):288-91. PMID 2009044
- [Background] Andrade Ortega JA, Delgado Martinez AD, Almecija Ruiz R. Validation of the Spanish version of the Neck Disability Index. Spine (Phila Pa 1976). 2010 Feb 15;35(4):E114-8. doi: 10.1097/BRS.0b013e3181afea5d. PMID 20110848
- [Background] Kovacs FM, Bago J, Royuela A, Seco J, Gimenez S, Muriel A, Abraira V, Martin JL, Pena JL, Gestoso M, Mufraggi N, Nunez M, Corcoll J, Gomez-Ochoa I, Ramirez MJ, Calvo E, Castillo MD, Marti D, Fuster S, Fernandez C, Gimeno N, Carballo A, Milan A, Vazquez D, Canellas M, Blanco R, Brieva P, Rueda MT, Alvarez L, Del Real MT, Ayerbe J, Gonzalez L, Ginel L, Ortega M, Bernal M, Bolado G, Vidal A, Ausin A, Ramon D, Mir MA, Tomas M, Zamora J, Cano A. Psychometric characteristics of the Spanish version of instruments to measure neck pain disability. BMC Musculoskelet Disord. 2008 Apr 9;9:42. doi: 10.1186/1471-2474-9-42. PMID 18400084
- [Background] Bahat HS, German D, Palomo G, Gold H, Nir YF. Self-Kinematic Training for Flight-Associated Neck Pain: a Randomized Controlled Trial. Aerosp Med Hum Perform. 2020 Oct 1;91(10):790-797. doi: 10.3357/AMHP.5546.2020. PMID 33187565
- [Background] Nagai T, Abt JP, Sell TC, Clark NC, Smalley BW, Wirt MD, Lephart SM. Neck proprioception, strength, flexibility, and posture in pilots with and without neck pain history. Aviat Space Environ Med. 2014 May;85(5):529-35. doi: 10.3357/asem.3874.2014. PMID 24834567
- [Background] Lopez-de-Uralde-Villanueva I, Notario-Perez R, Del Corral T, Ramos-Diaz B, Acuyo-Osorio M, La Touche R. Functional limitations and associated psychological factors in military personnel with chronic nonspecific neck pain with higher levels of kinesiophobia. Work. 2017;58(3):287-297. doi: 10.3233/WOR-172634. PMID 29154308
- [Background] Williams MA, McCarthy CJ, Chorti A, Cooke MW, Gates S. A systematic review of reliability and validity studies of methods for measuring active and passive cervical range of motion. J Manipulative Physiol Ther. 2010 Feb;33(2):138-55. doi: 10.1016/j.jmpt.2009.12.009. PMID 20170780
- [Background] Kauther MD, Piotrowski M, Hussmann B, Lendemans S, Wedemeyer C. Cervical range of motion and strength in 4,293 young male adults with chronic neck pain. Eur Spine J. 2012 Aug;21(8):1522-7. doi: 10.1007/s00586-012-2369-x. Epub 2012 May 17. PMID 22592882
- [Background] Lange B, Toft P, Myburgh C, Sjogaard G. Effect of targeted strength, endurance, and coordination exercise on neck and shoulder pain among fighter pilots: a randomized-controlled trial. Clin J Pain. 2013 Jan;29(1):50-9. doi: 10.1097/AJP.0b013e3182478678. PMID 23221624
- [Background] Simons DG. New views of myofascial trigger points: etiology and diagnosis. Arch Phys Med Rehabil. 2008 Jan;89(1):157-9. doi: 10.1016/j.apmr.2007.11.016. PMID 18164347
- [Background] Barbero M, Bertoli P, Cescon C, Macmillan F, Coutts F, Gatti R. Intra-rater reliability of an experienced physiotherapist in locating myofascial trigger points in upper trapezius muscle. J Man Manip Ther. 2012 Nov;20(4):171-7. doi: 10.1179/2042618612Y.0000000010. PMID 24179324
- [Background] Linde LD, Kumbhare DA, Joshi M, Srbely JZ. The Relationship between Rate of Algometer Application and Pain Pressure Threshold in the Assessment of Myofascial Trigger Point Sensitivity. Pain Pract. 2018 Feb;18(2):224-229. doi: 10.1111/papr.12597. Epub 2017 Jun 14. PMID 28440895
- [Background] Pousette MW, Lo Martire R, Linder J, Kristoffersson M, Ang BO. Neck Muscle Strain in Air Force Pilots Wearing Night Vision Goggles. Aerosp Med Hum Perform. 2016;87(11):928-932. doi: 10.3357/AMHP.4579.2016. PMID 27779951
- [Background] Ang B, Linder J, Harms-Ringdahl K. Neck strength and myoelectric fatigue in fighter and helicopter pilots with a history of neck pain. Aviat Space Environ Med. 2005 Apr;76(4):375-80. PMID 15828638
- [Background] Molina-Molina A, Ruiz-Malagon EJ, Carrillo-Perez F, Roche-Seruendo LE, Damas M, Banos O, Garcia-Pinillos F. Validation of mDurance, A Wearable Surface Electromyography System for Muscle Activity Assessment. Front Physiol. 2020 Nov 27;11:606287. doi: 10.3389/fphys.2020.606287. eCollection 2020. PMID 33329060
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Background] Calamita SAP, Biasotto-Gonzalez DA, De Melo NC, Fumagalli MA, Amorim CF, de Paula Gomes CAF, Politti F. Immediate Effect of Acupuncture on Electromyographic Activity of the Upper Trapezius Muscle and Pain in Patients With Nonspecific Neck Pain: A Randomized, Single-Blinded, Sham-Controlled, Crossover Study. J Manipulative Physiol Ther. 2018 Mar-Apr;41(3):208-217. doi: 10.1016/j.jmpt.2017.09.006. PMID 29549891
- [Background] Gomez-Perez L, Lopez-Martinez AE, Ruiz-Parraga GT. Psychometric Properties of the Spanish Version of the Tampa Scale for Kinesiophobia (TSK). J Pain. 2011 Apr;12(4):425-35. doi: 10.1016/j.jpain.2010.08.004. PMID 20926355
- [Background] Turner JA, Aaron LA. Pain-related catastrophizing: what is it? Clin J Pain. 2001 Mar;17(1):65-71. doi: 10.1097/00002508-200103000-00009. PMID 11289090
- [Background] Tascón M, Estevez R. La interacción entre la distracción y el catastrofismo en la respuesta al dolor. Jiménez A (ed): Comportamiento y palabra, 1a edición Estudios 2005 University, Málaga. 2005;119-21.
- [Background] Naranjo Orellana J, de la Cruz Torres B, Sarabia Cachadina E, de Hoyo M, Dominguez Cobo S. Two new indexes for the assessment of autonomic balance in elite soccer players. Int J Sports Physiol Perform. 2015 May;10(4):452-7. doi: 10.1123/ijspp.2014-0235. Epub 2014 Oct 29. PMID 25364865
- [Derived] Fernandez-Morales C, Espejo-Antunez L, Cardero-Duran MLA, Falla D, Moreno-Vazquez JM, Albornoz-Cabello M. Psychophysiological responses to a multimodal physiotherapy program in fighter pilots with flight-related neck pain: A pilot trial. PLoS One. 2024 Jul 5;19(7):e0306708. doi: 10.1371/journal.pone.0306708. eCollection 2024. PMID 38968243